CLINICAL TRIAL: NCT00001504
Title: A Phase I Trial of Tamoxifen and 9-Cis-Retinoic Acid in Breast Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 960080; 96-C-0080
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-01

CONDITIONS: Breast Cancer; Breast Neoplasm
Keywords: Retinoids; Biomarkers
MeSH Terms: conditions — Breast Neoplasms | interventions — Alitretinoin

INTERVENTIONS:
Drug: 9-cis-Retinoic Acid

SUMMARY:
This is a dosage escalation study to estimate the maximum tolerated dose of 9-cis-retinoic acid given in combination with tamoxifen. Groups of 3 to 6 patients receive oral 9-cis-retinoic acid daily for 4 weeks, after which daily oral tamoxifen is added to the regimen. Patients continue treatment for up to 28 weeks, with tamoxifen continued after the study if medically appropriate.

DETAILED DESCRIPTION:
This is a Phase I study of the combination tamoxifen and 9-cis-Retinoic acid in patients with breast cancer. The primary objective of the study is; 1) to determine the maximum tolerated dose of 9-cis-Retinoic acid in combination with Tamoxifen and to determine the overall and dose limiting toxicities. Other objectives are: 2) to determine the effect of Tamoxifen on the pharmacokinetics of 9-cis-Retinoic acid; 3) to evaluate the anti-tumor activity of this combination therapy within the context of a phase I study; 4) and to determine the expression of surrogate biomarkers of breast carcinogenesis before and after treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

All patients must have histologically documented diagnosis of Stage III, or IV breast carcinoma.

Patients with stage III that has completed chemotherapy: Estrogen receptor (ER) or progesterone receptor (PR) positive tumor required if premenopausal. Either ER/PR-positive or -negative tumor allowed if postmenopausal and have received prior chemotherapy.

Patients may have stage IV with ER/PR-positive or -negative tumor.

No CNS metastases, pseudotumor cereri, or seizures.

PRIOR/CONCURRENT THERAPY:

Patients who have ecovered from the toxic effects of prior therapy will be eligible.

Patients with prior tamoxifen will be allowed to participate. At least 3 weeks must have elapsed since the last dose of chemotherapy.

PATIENT CHARACTERISTICS:

Age: 18 and over.

Sex: Men and women.

Menopausal status: Any status.

Patients must have a performance status of ECOG 0-2.

Patients must have Hematopoietic criteria of:

ANC at least 1,500/mm(3).

Platelet count at least 90,000/mm(3).

Patients must have Hepatic criteria of:

In the absence of tumor involvement:

Bilirubin no greater than twice normal;

SGOT no greater than twice normal;

Alkaline phosphate no greater than twice normal;

Fasting triglycerides less than 3 times normal.

Patients must have Renal criteria of:

Serum creatinine no greater than 1.5 mg/dL OR;

Creatinine clearance at least 60 mL/min.

Other:

No allergy to study medications.

No nonmalignant systemic disease that would preclude therapy.

No second malignancy within 5 years except: Curatively treated basal cell skin carcinoma. Cervical carcinoma in situ.

Pregnant women will be excluded.

Negative pregnancy test required within 7 days prior to entry.

Adequate contraception required for 4 weeks prior to, during, and for 1 year after study.

Patients must give informed consent.

Patients who are poor medical or psychiatric risks will be eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18
Dates: Start 1996-05; Study Completion 2002-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Fontana JA. Interaction of retinoids and tamoxifen on the inhibition of human mammary carcinoma cell proliferation. Exp Cell Biol. 1987;55(3):136-44. doi: 10.1159/000163409. PMID 3666278
- [Background] Welsch CW, DeHoog JV. Retinoid feeding, hormone inhibition, and/or immune stimulation and the genesis of carcinogen-induced rat mammary carcinomas. Cancer Res. 1983 Feb;43(2):585-91. PMID 6401220
- [Background] Jordan VC, Murphy CS. Endocrine pharmacology of antiestrogens as antitumor agents. Endocr Rev. 1990 Nov;11(4):578-610. doi: 10.1210/edrv-11-4-578. No abstract available. PMID 2292243